CLINICAL TRIAL: NCT01753544
Title: Endoscopic Submucosal Dissection Using a Thulium Laser: Preliminary Results of a New Method for Treatment of Gastric Epithelial Neoplasia
Brief Title: Endoscopic Submucosal Dissection Using a Thulium Laser
Status: Completed | Type: Observational
Sponsor: Soonchunhyang University Hospital (Other)
Responsible Party: Principal Investigator, Jun-Hyung Cho, Clinical and Research Fellow, Soonchunhyang University Hospital
Other Study IDs: SCH-ESD-2012; NCT01838837 (obsolete NCT alias)
Record Dates: First submitted 2012-12-17; First posted 2012-12-20 (Estimated); Last update posted 2015-11-17 (Estimated); Status verified 2015-11

CONDITIONS: Gastric Dysplasia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — ESD specimen will be examined by a experienced pathologist.
Oversight: Data Monitoring Committee: Yes

SUMMARY:
We aim to evaluate safety and feasibility of a thulium laser system in performing endoscopic submucosal dissection of gastric neoplasia.

DETAILED DESCRIPTION:
Instead of endoscopic knives, a thin, flexible fiber is inserted through the working channel of the endoscope. Acetic acid (1.5%) and indigo carmine dye are sprayed onto the lesion to clarify the margin. Markings are made 10 mm outside the tumor margin using a laser fiber with a power setting at 30 W. After marking, a mixture of sodium hyaluronate with indigo carmine and epinephrine (1:25000) is injected into the submucosa outside the marking dots. A circumferential mucosal incision and submucosal dissection are performed by a thulium laser fiber with a power setting at 30 to 40 W. Activation of the laser beam is controlled by stepping on a foot pedal. Hemostasis during procedure is also attempted using the thulium laser. When hemostasis is not achieved properly, additional use of hemostatic forceps or a hemoclip will be considered.

ELIGIBILITY:
Inclusion Criteria:

* biopsy-proven gastric epithelial neoplasia

Exclusion Criteria:

* a.differentiated adenocarcinoma, ulcer(+), more than 3cm b.differentiated adenocarcinoma, submucosal invasion(+), more than 3cm c.undifferentiated adenocarcinoma, more than 2cm

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All patients are diagnosed with gastric epithelial neoplasia in a private clinic and referred to our hospital for endoscopic resection.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2012-10; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Technical success | 1 day
  Curative resection rate

SECONDARY OUTCOMES:
Complication rate | 7 days
  Procedure-related bleeding, perforation

CONTACTS AND LOCATIONS:
Overall Officials: Joo Young Cho, M.D., Principal Investigator — Digestive Disease Center, Soonchunhyang University Hospital
Locations (1):
- Digestive Disease Center, Soonchunhyang University Hospital, Seoul, South Korea

REFERENCES:
- [Background] Wendt-Nordahl G, Huckele S, Honeck P, Alken P, Knoll T, Michel MS, Hacker A. Systematic evaluation of a recently introduced 2-microm continuous-wave thulium laser for vaporesection of the prostate. J Endourol. 2008 May;22(5):1041-5. doi: 10.1089/end.2007.0421. PMID 18377234
- [Background] Xia SJ, Zhuo J, Sun XW, Han BM, Shao Y, Zhang YN. Thulium laser versus standard transurethral resection of the prostate: a randomized prospective trial. Eur Urol. 2008 Feb;53(2):382-89. doi: 10.1016/j.eururo.2007.05.019. Epub 2007 Jun 4. PMID 17566639
- [Background] Gotoda T, Yamamoto H, Soetikno RM. Endoscopic submucosal dissection of early gastric cancer. J Gastroenterol. 2006 Oct;41(10):929-42. doi: 10.1007/s00535-006-1954-3. Epub 2006 Nov 9. PMID 17096062
- [Background] Dray X, Donatelli G, Krishnamurty DM, Dubcenco E, Wroblewski RJ, Assumpcao L, Giday SA, Buscaglia JM, Shin EJ, Magno P, Pipitone LJ, Marohn MR, Kantsevoy SV, Kalloo AN. A 2-microm continuous-wave laser system for safe and high-precision dissection during NOTES procedures. Dig Dis Sci. 2010 Sep;55(9):2463-70. doi: 10.1007/s10620-010-1214-5. PMID 20704034